CLINICAL TRIAL: NCT07358000
Title: AIMSI Trial : Double-blind, Randomized, Non-inferiority Trial in Atopic Dermatitis: Comparison of Lipikar Balm and Relipid+ Balm in the Treatment of Mild to Moderate Atopic Dermatitis in Children and Adults
Brief Title: Double-blind, Randomized, Non-inferiority Trial in Atopic Dermatitis: Comparison of Lipikar Balm and Relipid+ Balm in the Treatment of Mild to Moderate Atopic Dermatitis in Children and Adults
Acronym: AIMSI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-A02369-38
Record Dates: First submitted 2025-06-19; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis; Emollients
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bras Lipikar AP+M (La Roche Posay) (Active Comparator)
  Interventions: Other: Baume Relipid+
- Bras baume RELIPID+ (Laboratoires Gilbert) (Experimental)
  Interventions: Other: Baume Relipid+

INTERVENTIONS:
Other: Baume Relipid+ — Application of daily emollient

SUMMARY:
The therapeutic cornerstone for mild to moderate forms of atopic dermatitis (AD) relies on the combination of topical corticosteroids and emollients. However, the daily application of emollients can be burdensome, leading to poor adherence, treatment fatigue, and therapeutic failure, often prompting a switch in emollient products.

Emollients therefore represent a true therapeutic challenge. They also raise economic concerns, as they are not reimbursed by national health insurance, unlike topical corticosteroids. This results in an out-of-pocket expense for patients, adding a significant financial burden in the context of this chronic skin condition.

Laboratoires Gilbert have developed and patented an active ingredient derived from seawater (Active Oligo Skin), formulated and produced at their pharmaceutical site in Hérouville Saint Clair. This active compound has shown promising in vitro and preclinical results in modulating inflammatory mechanisms involved in sensitive and atopic skin.

The objective of this clinical trial is to compare the efficacy of Laboratoires Gilbert's patented emollient balm (Relipid+) with a reference emollient balm considered the "gold standard" and most frequently prescribed on the market (Lipikar Baume AP+M, La Roche-Posay) for atopic dermatitis. The hypothesis is that the test balm will be at least as effective as the gold standard (non-inferiority) in clinical terms, with an added benefit on microbiome diversity-an emerging and critical issue in the management of atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 6 months to 70 years with mild to moderate atopic dermatitis (SCORAD < 40)

Time to treatment initiation < 72 hours between initial assessment and balm application

Affiliated with the French national health insurance system and French-speaking

Written informed consent must be obtained

Exclusion Criteria:

Patients who decline participation

Patients under legal guardianship, curatorship, legal protection, or judicial safeguard

Patients with a SCORAD indicating the need for systemic therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
SCORAD measurment | Day 0; Day 7; Day 28; Day 70
  SCORAD (Scoring Atopic Dermatitis) : from 0 up to 103

SECONDARY OUTCOMES:
DLQI (Quality of life) | Day 7 and Day 14
  DLQI questionnaire, scoring to 0 up to 30
Itch NRS scale (Itch Numeric Rating Scale) | Day 4 and Day 14
  Itch Numeric Rating Scale from 0 to 10
Use of topical steroids | Day 70 at the end of the study
  Amount of topical steroids used

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No